CLINICAL TRIAL: NCT06000891
Title: A Randomised, Multiple Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP7570 Administered in Subjects With Overweight or Obesity
Brief Title: A Trial Assessing Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP7570
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision by Sponsor; LSLV was completed on 21-Mar-2025 as planned.
Sponsor: Zealand Pharma (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP7570-23012; 2022-500614-26 (EudraCT Number)
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Safety and Tolerability
Keywords: GLP-1/GLP-2 agonist, overweight, obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The trial is a single-centre, randomised and double-blind within cohorts, placebo-controlled, sequential multiple ascending dose trial including three cohorts for Part 1 in a semi-parallel design and one cohort for Part 2.
Who Masked: Participant, Investigator
Masking Description: Unblinding for Part 1 will be performed after completion of Part 1 (cohort 1-3) of the trial. Everyone involved in the conduct of Part 2 of the trial will be blinded until completion of Part 2 (cohort 4) of the trial and the final data review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP7570 (Active Comparator): ZP7570 for subcutaneous once-weekly injection.
  Interventions: Drug: ZP7570
- Placebo (Placebo Comparator): Placebo for subcutaneous once-weekly injection. Corresponding volume matching active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP7570 — 13 once-weekly subcutaneous injections in Part 1. 28 once-weekly subcutaneous injections in Part 2.
  Other Names: GLP-1/GLP-2 agonist
  Arms: ZP7570
Drug: Placebo — 13 once-weekly subcutaneous injections in Part 1. 28 once-weekly subcutaneous injections in Part 2.
  Arms: Placebo

SUMMARY:
The trial is a Phase 1, single-centre, randomised and double-blind within cohorts, placebo-controlled, sequential multiple ascending dose trial including three cohorts in Part 1 in a semi-parallel design and one cohort in Part 2 in overweight and obese but otherwise healthy subjects, randomised to ZP7570 or placebo within each cohort where the observational period is 18 weeks for Part 1 and 28 weeks for Part 2. All subjects will be dosed for 13 weeks in Part 1 and for 28 weeks in Part 2 with ascending weekly doses of ZP7570 at dose levels with corresponding volume of placebo.

DETAILED DESCRIPTION:
ZP7570 is a dual GLP-1R/GLP-2R agonist in clinical development for weight management. The overall purpose of this trial is to evaluate the safety and tolerability when applying dose titration of ascending doses of ZP7570 and at steady state.

The trial is a Phase 1, single-centre, randomised and double-blind within cohorts, placebo-controlled, sequential multiple ascending dose trial including three cohorts in Part 1 in a semi-parallel design and one cohort in Part 2 in overweight and obese but otherwise healthy subjects, randomised to ZP7570 or placebo. All subjects will be dosed with ascending weekly doses of ZP7570 with corresponding volume of placebo. After informed consent has been obtained, eligibility of the subjects will be assessed during a screening Visit (V1). Additional tests to assess safety and PK and PD will take place during in-house visits and ambulatory visits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years, both inclusive.
* Body Mass Index (BMI) between 27.0 and 39.9 kg/m^2, both inclusive.
* In overall good health according to age (medical history, physical and neurological examination, vital signs, and laboratory assessments), as judged by the investigator at screening.

Exclusion Criteria:

* History of gastrointestinal (GI) diseases including functional complaints that could interfere with the pharmacokinetics of the IMP or auxiliary medicinal product (acetaminophen) of the trial.
* Any relevant abnormal renal parameters in the following ranges:

Serum creatinine above UNL+10% or normalised estimated glomerular filtration rate (eGFR) below 60.0 l/min/1.73m2, as defined by CKD-EPI.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 2. Male subject or female subject of non-child-bearing potential A woman is considered of childbearing potential following menarche and until becoming postmenopausal unless permanently sterile due to hysterectomy, or bilateral salpingectomy, or bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
Enrollment: 84 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Day 1 to Day 127 in Part 1. Day 1 to Day 232 in Part 2
  Incidence of treatment emergent adverse events (TEAEs) from first dose (Day 1) to end of trial (Day 127) in Part 1.
  Incidence of treatment emergent adverse events (TEAEs) from first dose (Day 1) to end of trial (Day 232) in Part 2.

SECONDARY OUTCOMES:
Pharmacokinetics endpoints related to ZP7570 exposure | Area under the drug concentration curve from baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics: Area under the plasma concentration curve from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics: Area under the plasma concentration curve from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Maximum drug concentration (Cmax) from baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Maximum plasma concentration (peak) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Maximum plasma concentration (peak) from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Time to maximum plasma concentration from baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Time to maximum plasma concentration (Tmax) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Time to maximum plasma concentration (Tmax) from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Elimination rate constant from baseline baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Elimination rate constant (λz) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Elimination rate constant (λz) from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Elimination half-life from baseline baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Elimination half-life (t1/2) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Elimination half-life (t1/2) from baseline (Day 1, predose) to 22 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Apparent volume of distribution from baseline baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Apparent volume of distribution (Vz/f) during the terminal phase from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Apparent volume of distribution (Vz/f) during the terminal phase from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Apparent total clearance of the drug from plasma from baseline baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.)
  Pharmacokinetics - Apparent total clearance of the drug from plasma (Cl/f) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Apparent total clearance of the drug from plasma (Cl/f) from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Pharmacokinetics endpoints related to ZP7570 exposure | Trough concentration measured from baseline baseline (Day 1) to 18 weeks (Day 127) in Part 1 and to 33 weeks (Day 232) in Part 2.
  Pharmacokinetics - Trough concentration measured predose (Ctrough) from baseline (Day 1, predose) to 18 weeks (Day 127) in Part 1.
  Pharmacokinetics - Trough concentration measured predose (Ctrough) from baseline (Day 1, predose) to 33 weeks (Day 232) in Part 2.
Absolute change in body weight | Day 1 and Day 92 in Part 1. Day 1 and Day 197 in Part 2.
  Absolute change in body weight in kilogram (kg) from baseline (Day 1) to end of treatment (Day 92) in Part 1.
  Absolute change in body weight in kilogram (kg) from baseline (Day 1) to end of treatment (Day 197) in Part 2.
Percent change in body weight | Day 1 and Day 92 in Part 1. Day 1 and Day 197 in Part 2.
  Percent change in body weight in percent (%) from baseline (Day 1) to end of treatment (Day 92) in Part 1.
  Percent change in body weight in percent (%) from baseline (Day 1) to end of treatment (Day 197) in Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hoevelmann, MD, Principal Investigator — Profil, Neuss, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The data collection and handling of clinical trial data at the trial site has been designed to limit the possibility of identifying trial subjects from their data. To this end, pseudonymised data will be used wherever possible and the collection of demographic information that could be used for re-identification of subjects will be restricted to the extent necessary for the conduct of this trial.